CLINICAL TRIAL: NCT00073476
Title: A Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of a 72-Hour Infusion of CP-101,606 in Subjects With Acute Ischemic Stroke.
Brief Title: A Study to Evaluate the Efficacy and Safety of CP-101,606 in Subjects With an Acute Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1611005
Record Dates: First submitted 2003-11-21; First posted 2003-11-24 (Estimated); Last update posted 2006-06-22 (Estimated); Status verified 2006-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — traxoprodil mesylate

INTERVENTIONS:
Drug: traxiprodil (CP-101,606)

SUMMARY:
The purpose of this study is to determine whether a new research medication is effective and safe for the treatment of acute stroke when given within 6 hours of the onset of stroke.

ELIGIBILITY:
Inclusion Criteria:

Males & females age 40-90 years

Enrolled in study within 6 hours of onset of stroke symptoms

Willing to sign informed consent form

No significant disabilities prior to stroke

Exclusion Criteria:

Treatment with t-PA (tissue plasminogen activator)

Premorbid modified rankin scale score of 2 or more

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-09; Study Completion 2005-02

PRIMARY OUTCOMES:
No or minimal neurological deficit at last visit
Marked neurological improvement at last visit

SECONDARY OUTCOMES:
Modified Rankin scale at last visit
Mortality
Safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (8):
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
- Pfizer Investigational Site, Tartu, Estonia
- Germany (4):
  - Pfizer Investigational Site, Bad Neustadt an der Saale
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Lübeck
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Győr
- Italy (2):
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Perugia
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Pfizer Investigational Site, Singapore, Singapore
- Spain (3):
  - Pfizer Investigational Site, Santiago de Compostela, Galicia
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Zaragoza

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1611005&StudyName=A+Study+to+Evaluate+the+Efficacy+and+Safety+of++CP%2D101%2C606+in+Subjects+With+an+Acute+Stroke+